CLINICAL TRIAL: NCT07173166
Title: Randomized, Multicenter, Controlled Clinical Trial to Evaluate the Efficacy of Non-Pharmacological Interventions on Neurotoxicity Associated With CAR-T Therapy in Hematologic Patients
Brief Title: Non-Pharmacological Interventions for Neurotoxicity in Hematologic Patients Receiving CAR-T Therapy
Acronym: CARE-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Marina Hernández Aliaga, Principal Investigator, Instituto de Investigacion Sanitaria INCLIVA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/185
Record Dates: First submitted 2025-08-16; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Cancer
Keywords: CAR-T therapy; Neurotoxicity; Nutrition; Physical activity
MeSH Terms: conditions — Hematologic Neoplasms; Neurotoxicity Syndromes; Motor Activity | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The intervention is assigned and administered by external staff. Investigators do not participate in delivering the interventions. Outcome assessors are also blinded. Participants are aware of their assigned intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity (Experimental): Patients assigned to intervention group A will follow a supervised programme of physical activity and exercise at home and during their hospital stay. These recommendations are designed and supervised by a physiotherapist. The programme will include three weekly aerobic exercise sessions and two resistance exercise sessions, as recommended in the literature. Each session will last approximately 35 minutes and will include a warm-up, training and cool-down.
  All patients will follow the same exercise programme, which will be adapted to a basic, intermediate and advanced level to adapt to the patients' physical condition. The loads, intensity and number of sets will be adapted for each level.
  The programme is scheduled to commence one month prior to the initiation of CAR-T therapy. It is recommended that patients adhere to the professional's guidelines for a period of at least one month following treatment.
  Interventions: Other: Physical activity
- Physical activity and nutrition (Experimental): The intervention combines a structured physical activity programme with individualised nutritional recommendations based on the Mediterranean diet. These recommendations are designed and supervised by a nutritionist and a physiotherapist. The macronutrient distribution followed standard guidelines (50-55% carbohydrates, 30-35% fats, 10-15% proteins), emphasising vegetables, fruits, legumes, cereals, dairy, lean meats, fish, nuts, and olive oil. Each food group contributes bioactive compounds with anti-inflammatory and antioxidant properties, including lycopene, quercetin, anthocyanins, genistein, ferulic acid, SCFAs, omega-3 fatty acids and polyphenols. These have been shown to mitigate oxidative stress, inflammation and toxicological effects, thereby supporting cardio.
  The programme is scheduled to commence one month prior to the initiation of CAR-T therapy. It is recommended that patients adhere to the professional's guidelines for a period of at least one month following treatment.
  Interventions: Other: Physical activity; Other: Physical activity and nutrition
- Control (No Intervention): The control group will serve to establish a baseline for identifying clinical, demographic, and response patterns of the studied variables. All procedures and interventions will be conducted in accordance with the center's standard clinical practice.

INTERVENTIONS:
Other: Physical activity — Patients assigned to intervention group A will follow a supervised programme of physical activity and exercise at home and during hospitalisation. All patients will follow the same exercise programme, which will be adapted to a basic, intermediate and advanced level to suit the patients' physical condition. The loads, intensity and number of sets will be adapted to each level.
  Aerobic exercise will consist of walking and/or cycling at an intensity of between two and five on the Borg perceived exertion (RPE) scale. Resistance exercise will consist of one session focusing on the trunk and upper limbs, and another on the lower limbs. Both sessions will include seven exercises, performed at an intensity of between three and four on the Borg RPE scale.
  Arms: Physical activity; Physical activity and nutrition
Other: Physical activity and nutrition — The intervention integrates a structured physical activity programme with individualized nutritional recommendations based on the Mediterranean diet. Macronutrient distribution was 50-55% carbohydrates, 30-35% fats, and 10-15% proteins. The protocol emphasized the intake of vegetables (≥2 servings/day, 200 g each), fruits (1-2 servings/day, 150 g each), legumes (≥3 servings/week, 150 g cooked), whole grains (1-2 servings/meal, 40-60 g), and low-fat dairy products (1-2 servings/day; 200 ml milk or 125 g yoghurt). Lean meats were prescribed at 3-4 servings/week (100-125 g each), fish and seafood at 4 servings/week (150 g each), nuts at 3-7 servings/week (30 g each), and olive oil as the principal fat source (≤4 tbsp/day). Micronutrients and bioactive compounds from these foods, including antioxidants, polyphenols, and essential fatty acids, were recognized as pivotal for modulating protective mechanisms and mitigating toxicological effects.
  Arms: Physical activity and nutrition

SUMMARY:
The goal of this clinical trial is to learn if two non-pharmacological strategies can help reduce neurotoxicity caused by CAR-T cell therapy in adult patients with hematologic cancer, both sexes, aged 18 to 80 years. The strategies are:

* A structured physical activity program.
* A combination of physical activity and nutritional recommendations.

The main questions it aims to answer are:

* Does physical activity help lower the risk or severity of neurotoxicity after CAR-T therapy?
* Does combining physical activity with nutritional recommendations provide greater protection against neurotoxicity than physical activity alone?

Researchers will compare two intervention groups with a control group (no intervention) to see which approach is most effective in reducing neurotoxicity and improving recovery.

Participants will be randomly assigned to one of three groups using stratified randomization to ensure balanced clinical and demographic characteristics:

* Group A: Structured physical activity program.
* Group B: Structured physical activity program combined wuth nutritional recommendations.
* Group C: No intervention; used to establish baseline patterns.

Participants will be evaluated periodically by study professionals. Comprehensive records of symptoms, health measurements, and relevant lifestyle data will be maintained throughout the study.

DETAILED DESCRIPTION:
A parallel-group, multicenter and randomized controlled clinical trial will be conducted from July 2025 to July 2027. The study will evaluate the effectiveness of two non-pharmacological interventions in reducing neurotoxicity associated with CAR-T cell therapy in adult patients with hematologic cancer.

A total of 100 patients will be enrolled and randomly assigned into three groups using stratified randomization performed by an individual external to the research team.

The intervention will begin at least one month prior to CAR-T cell infusion. Participants will be followed weekly before, during, and for four weeks after therapy. Interventions and evaluations will be carried out in the same hospital where the patient receives treatment, and always by the same multidisciplinary team (hematologists, nurses, nutritionists, physiotherapists).

Primary and secondary outcomes will be assessed at baseline (prior to intervention), during treatment, and post-treatment follow-up. Written informed consent will be obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18 to 80 years.
* Diagnosed with a hematological condition.
* Initiating antineoplastic treatment with CAR-T cell therapy.

Exclusion Criteria:

* Presence of language barriers or physical and/or cognitive impairments that hinder the understanding of the interventions or prevent proper completion of the assessment tools used in the study.
* Pre-existing neurological or psychiatric comorbidities that may interfere with the evaluation of neurotoxic effects of the hematologic treatment.
* Concomitant treatment with additional neurotoxic drugs not related to the study protocol.
* History of abusive consumption of neurotoxic substances.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of neurotoxicity as assessed by CTCAE v5.0 and Immune Effector Cell-Associated Encephalopathy (ICE) score following CAR-T therapy | At baseline and from the infusion of treatment until 6 months after CAR-T therapy.
  Patients will undergo a standardised neurological assessment. Neurotoxicity will be graded according to version 5.0 of the Common Terminology Criteria for Adverse Events (CTCAE). The Immune Effector Cell-Associated Encephalopathy (ICE) score will also be used to evaluate five cognitive domains, for which the maximum possible score is 10. The following will be assessed: orientation (year, month, city, hospital; 4 points); object naming (three objects; 3 points); following commands (two-step command; 1 point); writing a coherent sentence (1 point); and attention (counting backwards from 100 in tens; 1 point). Lower ICE scores reflect greater neurological impairment.

SECONDARY OUTCOMES:
Functional independence as assessed by the Lawton and Brody Instrumental Activities of Daily Living (IADL) scale | At baseline and from the infusion of treatment until 6 months after CAR-T therapy.
  Functional capacity will be assessed using the Lawton and Brody Instrumental Activities of Daily Living (IADL) scale . This instrument evaluates the patient's ability to perform eight instrumental activities essential for independent living (e.g., using the telephone, shopping, preparing meals, housekeeping, laundry, transportation, medication management, and financial management). Each item is scored as 0 (dependent) or 1 (independent), yielding a total score ranging from 0 (total dependence) to 8 (complete independence). Higher scores indicate greater independence and better functional status.
Physical activity level as assessed by the International Physical Activity Questionnaire (IPAQ) | At baseline and from the infusion of treatment until 6 months after CAR-T therapy.
  Physical activity will be quantified using the International Physical Activity Questionnaire (IPAQ). The instrument comprises seven items and provides information on the time spent walking, performing moderate-intensity activities, vigorous-intensity activities, and sedentary behaviour during the last seven days. The results are expressed in metabolic equivalent task minutes per week (MET-min/week) and categorised into three levels of physical activity:
  * Low: no or insufficient activity.
  * Moderate: ≥3 days of vigorous activity (20 minutes/day), ≥5 days of moderate activity or walking (30 minutes/day), or a combination reaching ≥600 MET-min/week.
  * High: vigorous activity on ≥3 days achieving ≥1,500 MET-min/week, or 7 days of any combination reaching ≥3,000 MET-min/week.
  This classification allows the identification of patients at risk of inactivity and facilitates monitoring of changes across the intervention.
Nutritional status as assessed by the Patient-Generated Subjective Global Assessment (PG-SGA) | At baseline and from the infusion of treatment until 6 months after CAR-T therapy.
  Nutritional status will be evaluated using the Patient-Generated Subjective Global Assessment (PG-SGA), a tool that has been validated for the purpose of nutritional screening in oncohematology. The PG-SGA combines patient-reported data and clinician assessment, including weight changes, dietary intake, nutrition impact symptoms, functional capacity, and physical examination findings. Patients are categorised into three groups: well-nourished, moderately malnourished/at risk of malnutrition, or severely malnourished. The instrument facilitates the identification of patients requiring nutritional interventions, thereby providing a comprehensive overview of nutritional risk within the study population.
Quality of life as assessed by the Short Form 12 (SF-12) | At baseline and from the infusion of treatment until 6 months after CAR-T therapy.
  Quality of life will be assessed using the Short Form 12 (SF-12) health survey. The SF-12 evaluates eight health domains, which are aggregated into two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Each domain is scored according to the SF-12 scoring algorithm, resulting in standardized scores ranging from 0 to 100, with higher scores indicating better health-related quality of life.
Adherence to interventions | At baseline and from the infusion of treatment until 6 month after CAR-T therapy.
  The researcher collected attendance records, food records and self-reported activity levels as part of the follow-up of the subjects.

OTHER OUTCOMES:
Length of initial hospital stay | From the infusion of treatment until 6 months after CAR-T therapy.
  Duration of the initial hospitalisation following CAR-T infusion will be documented from the day of admission until discharge (days).
Number of hospital readmissions | From the infusion of treatment until 6 months after CAR-T therapy.
  Hospital readmissions related to the intervention will be documented, including cause and date of readmission (number of readmissions per participant).

CONTACTS AND LOCATIONS:
Overall Officials: Marina Hernandez Aliaga, RN, MSc, PhD(c), Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA
Locations (2):
- Spain (2):
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
The dissemination of individual participant data will not occur directly. All information related to the study, including the protocol, detailed study design, primary and secondary outcomes, and summary results, will be shared through peer-reviewed scientific publications, conference abstracts, and academic presentations. This approach ensures full transparency of the study's methodology, analyses, and findings, while strictly protecting participant privacy, maintaining confidentiality, and complying with all relevant ethical, legal, and regulatory standards.

REFERENCES:
- [Background] Borsati A, Murri A, Natalucci V, Cerulli C, Barbieri E, Lucertini F, Lanza M, Parisi A, Galvani C, Buono P, Mancini A, Fischetti F, Poli L, Di Blasio A, Iannaccone A, Avancini A, Mauri C, Ferri Marini C, Grazioli E. The Effect of Exercise-Based Interventions on Health-Related Quality of Life of Patients with Hematological Malignancies: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2025 Feb 21;13(5):467. doi: 10.3390/healthcare13050467. PMID 40077029
- [Background] Richards J, Arensberg MB, Thomas S, Kerr KW, Hegazi R, Bastasch M. Impact of Early Incorporation of Nutrition Interventions as a Component of Cancer Therapy in Adults: A Review. Nutrients. 2020 Nov 5;12(11):3403. doi: 10.3390/nu12113403. PMID 33167544
- [Background] Hayden PJ, Roddie C, Bader P, Basak GW, Bonig H, Bonini C, Chabannon C, Ciceri F, Corbacioglu S, Ellard R, Sanchez-Guijo F, Jager U, Hildebrandt M, Hudecek M, Kersten MJ, Kohl U, Kuball J, Mielke S, Mohty M, Murray J, Nagler A, Rees J, Rioufol C, Saccardi R, Snowden JA, Styczynski J, Subklewe M, Thieblemont C, Topp M, Ispizua AU, Chen D, Vrhovac R, Gribben JG, Kroger N, Einsele H, Yakoub-Agha I. Management of adults and children receiving CAR T-cell therapy: 2021 best practice recommendations of the European Society for Blood and Marrow Transplantation (EBMT) and the Joint Accreditation Committee of ISCT and EBMT (JACIE) and the European Haematology Association (EHA). Ann Oncol. 2022 Mar;33(3):259-275. doi: 10.1016/j.annonc.2021.12.003. Epub 2021 Dec 16. PMID 34923107
- [Background] Han MW, Jeong SY, Suh CH, Park H, Guenette JP, Huang RY, Kim KW, Yoon DH. Incidence of immune effector cell-associated neurotoxicity among patients treated with CAR T-cell therapy for hematologic malignancies: systematic review and meta-analysis. Front Neurol. 2024 Oct 15;15:1392831. doi: 10.3389/fneur.2024.1392831. eCollection 2024. PMID 39474369